CLINICAL TRIAL: NCT01066247
Title: The Influence of HRV-changing Premedication on Hemodynamic Parameters After Spinal Anesthesia
Brief Title: Premedication and Haemodynamics After Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Dr Radoslaw Owczuk, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GUMed-Ow-001
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2010-01

CONDITIONS: Hemodynamics After Spinal Anesthesia
Keywords: spinal anesthesia; heart rate variability; premedication; heart rate; blood pressure
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Active Comparator): intramuscular midazolam 15 mg given 30 minutes before spinal blockade performing
  Interventions: Drug: Midazolam
- Morphine (Active Comparator): intramuscular morphine 10 mg given 30 minutes before spinal blockade performing
  Interventions: Drug: Morphine hydrochloride; Midazolam

INTERVENTIONS:
Drug: Morphine hydrochloride; Midazolam — intramuscular morphine 10 mg given 30 minutes before spinal blockade performing
  Arms: Morphine
Drug: Midazolam — intramuscular midazolam 15 mg given 30 minutes before spinal blockade performing
  Arms: Midazolam

SUMMARY:
Blood pressure drop following spinal anesthesia is connected with sympathetic/parasympathetic activity which may be determinated by Heart Rate Variability (HRV) assessment. Sympathetic predomination expressed as LF/HF ratio above 2.5 is strongly connected with deeper blood pressure fall. As drugs given for premedication may have impact on HRV variables, the investigators would like to determine if pharmacological premedication may modify hemodynamic changes following spinal blockade. Two drugs will be compared - midazolam which is known to lead to increase in LF/HF ratio and morphine - opioid which provokes opposite effect.

ELIGIBILITY:
Inclusion Criteria:

* spinal blockade for elective surgery

Exclusion Criteria:

* contraindications for spinal anesthesia
* hypertension
* heart failure
* chronic respiratory failure
* hypersensitivity for midazolam or morphine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
hemodynamics after spinal anesthesia | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw Owczuk, Ph.D., Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland

REFERENCES:
- [Result] Hanss R, Renner J, Ilies C, Moikow L, Buell O, Steinfath M, Scholz J, Bein B. Does heart rate variability predict hypotension and bradycardia after induction of general anaesthesia in high risk cardiovascular patients? Anaesthesia. 2008 Feb;63(2):129-35. doi: 10.1111/j.1365-2044.2007.05321.x. PMID 18211442
- [Result] Hanss R, Bein B, Francksen H, Scherkl W, Bauer M, Doerges V, Steinfath M, Scholz J, Tonner PH. Heart rate variability-guided prophylactic treatment of severe hypotension after subarachnoid block for elective cesarean delivery. Anesthesiology. 2006 Apr;104(4):635-43. doi: 10.1097/00000542-200604000-00005. PMID 16571956
- [Result] Owczuk R, Wenski W, Polak-Krzeminska A, Twardowski P, Arszulowicz R, Dylczyk-Sommer A, Wujtewicz MA, Sawicka W, Morzuch E, Smietanski M, Wujtewicz M. Ondansetron given intravenously attenuates arterial blood pressure drop due to spinal anesthesia: a double-blind, placebo-controlled study. Reg Anesth Pain Med. 2008 Jul-Aug;33(4):332-9. doi: 10.1016/j.rapm.2008.01.010. PMID 18675744
- [Result] Hidaka S, Kawamoto M, Kurita S, Yuge O. Comparison of the effects of propofol and midazolam on the cardiovascular autonomic nervous system during combined spinal and epidural anesthesia. J Clin Anesth. 2005 Feb;17(1):36-43. doi: 10.1016/j.jclinane.2004.03.012. PMID 15721728